CLINICAL TRIAL: NCT01693913
Title: Effects of a Cognitive-behavioral Weight Loss Treatment
Brief Title: Cognitive-behavioral Weight Loss Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approval canceled
Sponsor: YMCA of Metropolitan Atlanta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YMCAAtlantaWeightLoss
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Weight
MeSH Terms: conditions — Body Weight | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-behavioral (Experimental): Those participating in a cognitive behaviorally supported exercise and nutrition treatment will receive a cognitive behavioral exercise and nutrition over 50 weeks
  Interventions: Behavioral: cognitive behavioral exercise and nutrition over
- Nurtition education (Active Comparator): This arm will participate in nutrition and exercise education
  Interventions: Behavioral: nutrition and exercise education

INTERVENTIONS:
Behavioral: cognitive behavioral exercise and nutrition over
  Arms: Cognitive-behavioral
Behavioral: nutrition and exercise education
  Arms: Nurtition education

SUMMARY:
That a treatment using a cognitive-behavioral treatment for exercise and nutrition support will be associated with greater weight loss that a treatment of nutrition and exercise education.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 21-60
* Body mass index 30-40 kg/m2

Exclusion Criteria:

* Pregnancy
* Medications for a psychological disorder
* Contraindications for exercise

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
weight | baseline, months 3,6,12, 24
  Direct measurement of weight

CONTACTS AND LOCATIONS:
Overall Officials: James J Annesi, PhD, Principal Investigator — YMCA of Metro Atlanta
Locations (1):
- YMCA of Metro Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Annesi JJ. Supported exercise improves controlled eating and weight through its effects on psychosocial factors: extending a systematic research program toward treatment development. Perm J. 2012 Winter;16(1):7-18. doi: 10.7812/11-136. PMID 22529754
- [Background] Annesi JJ, Marti CN. Path analysis of exercise treatment-induced changes in psychological factors leading to weight loss. Psychol Health. 2011 Aug;26(8):1081-98. doi: 10.1080/08870446.2010.534167. Epub 2011 Jul 25. PMID 21780982
- [Background] Annesi JJ, Unruh JL, Marti CN, Gorjala S, Tennant G. Effects of the coach approach intervention on adherence to exercise in obese women: assessing mediation of social cognitive theory factors. Res Q Exerc Sport. 2011 Mar;82(1):99-108. doi: 10.1080/02701367.2011.10599726. PMID 21462690